CLINICAL TRIAL: NCT02196792
Title: Assessment of Polyethylene Wear, Migration and Clinical Outcome in Total Hip Replacement - A Prospective Randomized Control Trial
Brief Title: Assessment of Polyethylene Wear, Migration and Clinical Outcome in Total Hip Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Abdalla Nommesen El-Sahoury, Research assistant, Odense University Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: project-ID S-20080151
Record Dates: First submitted 2014-07-14; First posted 2014-07-22 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis
Keywords: Joint Diseases; Musculoskeletal Diseases; radiostereometric analysis; Total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- E-Poly/32 mm (Active Comparator): E-Poly polyethylene liner in a titanium cup with a stem with 32 mm cobalt-chromium (CoCr) femoral head.
  Interventions: Device: E-Poly liner; Device: 32 mm femoral head
- E-Poly/36 mm (Active Comparator): E-Poly polyethylene liner in a titanium cup with a stem with 36 mm CoCr femoral head.
  Interventions: Device: E-Poly liner; Device: 36 mm femoral head
- ArComXL/32 mm (Active Comparator): ArComXL polyethylene liner in a titanium cup with a stem with 32 mm CoCr femoral head.
  Interventions: Device: ArComXL liner; Device: 32 mm femoral head
- ArComXL/36 mm (Active Comparator): ArComXL polyethylene liner in a titanium cup with a stem with 36 mm CoCr femoral head.
  Interventions: Device: ArComXL liner; Device: 36 mm femoral head

INTERVENTIONS:
Device: E-Poly liner — E-Poly liner with a titanium cup
  Arms: E-Poly/32 mm; E-Poly/36 mm
Device: ArComXL liner — ArComXL liner with a titanium cup
  Arms: ArComXL/32 mm; ArComXL/36 mm
Device: 32 mm femoral head — Stem with a 32 mm CoCr femoral head
  Arms: ArComXL/32 mm; E-Poly/32 mm
Device: 36 mm femoral head — Stem with a 36 mm CoCr femoral head
  Arms: ArComXL/36 mm; E-Poly/36 mm

SUMMARY:
The objective of the study is to investigate head penetration, cup migration, and clinical outcome in total hip replacements using a factorial design. Treatment groups are E-Poly versus ArComXL liners, and 36 mm versus 32 mm head size.

ELIGIBILITY:
Inclusion Criteria:

* Primary idiopathic arthritis,
* Eligible for uncemented total hip arthroplasty
* 40 to70 years of age,
* Cup size of 54mm and above

Exclusion Criteria:

* Anteversion where non-standard stem can be used,
* Dysplasia (Center-edge angle of Wiberg < 20°),
* Malignant condition
* Prior radiotherapy
* Physical or psychological condition that renders it impossible for the patient to take part in our usual rehabilitation programme (as stated in the department's standard operation procedure),
* Complications during surgery (requiring screws in shell or femoral cerclage)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-05-01; Primary Completion 2015-05-01 (Actual); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean head penetration from baseline to 5 year follow-up | From baseline to 5 years
  Mean head penetration assessed using röntgen steregrammetry analysis (RSA) from baseline to 5 year follow-up

SECONDARY OUTCOMES:
Mean cup migration form baseline to 5 year follow-up | From baseline to 5 years
  Mean cup migration assessed using RSA from baseline to 5 year follow-up
Mean change in clinical outcome score from baseline to 5 year follow-up | From baseline to 5 years
  Mean change in patient-reported hip function (Harris Hip Score), quality of life (EQ-5D and SF-36), and patient activity (UCLA Activity Score).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Abdalla N. El-Sahoury, BSc.med, Principal Investigator — OUH Den Ortopædkirurgiske Forskningsenhed; Ming Ding, Professor MD, Study Director — Odense University Hospital, University of Southern Denmark
Locations (1):
- Joseph Abdalla Nommesen El-Sahoury, Odense C, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT02196792/SAP_000.pdf